CLINICAL TRIAL: NCT05503680
Title: The Effect of a Yoga Intervention for Reducing Stress Among People Living With HIV in Indonesia: A Randomized Controlled Trial
Brief Title: The Effect of Yoga for Stress Among HIV Patients in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Jufri Hidayat, Principal investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2564/VII/SP/2022
Record Dates: First submitted 2022-07-22; First posted 2022-08-17 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: yoga; Stress, Psychological; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stress, Psychological | interventions — Yoga

STUDY DESIGN:
Masking Description: In this study, we will blind the data collector
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): The experimental group is people living with HIV who will receive 120 minutes per week of yoga intervention.
  Interventions: Behavioral: Yoga
- Control group (No Intervention): In this study, the control group will receive standard care where participants usually receive various program from The local HIV clinic including general education program, health check-up, and oral antiretroviral regimen

INTERVENTIONS:
Behavioral: Yoga — In this study, the researcher will provide participants with two month of Hatha yoga as an experimental intervention for managing stress. All participants who belong to the intervention group will be required to complete 120 minutes per week of home-based, online streaming yoga for eight weeks with our certified yoga instructor. The intervention will be conducted online by Zoom video; participants will be sent a link to join a scheduled live online yoga session twice every week. The data collection will be undertaken in three times: baseline (before the intervention begins), posttest one ( after two month intervention), and posttest two (one month after yoga intervention finish) to evaluate the lasting effect of yoga.
  Other Names: Hatha yoga
  Arms: Yoga group

SUMMARY:
This study is aimed to evaluate the effects of yoga intervention versus usual care (control group) for reducing stress among people living with HIV in Indonesia.

DETAILED DESCRIPTION:
Introduction: Human immunodeficiency virus (HIV) continues to be a public health challenge for four decades after the disease appeared. Stress is one of the most common mental health problems that occur among people living with HIV. Yoga is increasingly popular as one of the complementary therapies in health care systems including in nursing. Moreover, much evidence shows that yoga is a promising modality to be used to treat stress and to maintain the health and wellbeing of PLWH.

Purpose: The primary objective in this study is to evaluate the effects of yoga intervention versus usual care (control group) for reducing stress among people living with HIV in Indonesia.

Methods: This study will use a parallel group randomized controlled trial (RCT) design, with single blinding, and repeated measures. Sample will be divided into a yoga intervention group and a routine care group as the control group. In this study, the independent variable is defined as yoga intervention, and the dependent variable is stress. In total, participants who will participate is sixty-six, thirty-three participants in yoga group and thirty-three in control group. The Generalized Estimating Equation will be performed for the data analysis.

ELIGIBILITY:
Inclusion Criteria:

Participants are patients who

* Had been diagnosed with HIV.
* Were newly diagnosed or had taken ARV medication for at least one month.
* Are age 18 years or older.
* Have access to a desktop, laptop, or smartphone on a regular basis.
* Have access to reliable internet.
* Are fluent in Indonesian.
* Are willing to participate and sign the consent form.
* Are willing to be blood tested for CD4 counts or viral load at baseline and eight weeks after the intervention.

Exclusion Criteria:

Patients who did not qualify to participate were:

* Those who reported performing yoga or other body-mind exercises at least one-month prior to the start of this study.
* Those who were not in physically fit condition
* Those who had been diagnosed with musculoskeletal problems, i.e., osteoporosis, osteoarthritis, bone injury, or spine problems.
* Those who have difficulty keeping their balance.
* Those who are currently pregnant, or plan to become pregnant during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Perceived stress scale (this study will measure the the phenomenon of stress among PLWH using the Perceived Stress Scale developed by Dr. Sheldon Cohen in 1983). | (1) Pre-test (before yoga intervention), (2) Post-test one / at the week-eight (after yoga intervention finish), (3) Post-test two for following up (at the week twelve or one month after yoga intervention finish).
  The scale uses a 5-point rating scale from never (0) to very often (4) to measure the degree to which a person judges situations in their life to be stressful. This scale contains 10 items. Scores range from 1 to 40, with higher scores reflecting greater perceived stress. This scale has sufficient internal consistency with Cronbach alpha 0.78 (Cohen et al., 1983). The stress will be measured in three different time to see how the yoga intervention change the level of stress of participants, before and after intervention.

SECONDARY OUTCOMES:
The Brief Health status Survey | (1) Pre-test (before yoga intervention), (2) Post-test one / at the week-eight (after yoga intervention finish), (3) Post-test two for following up (at the week twelve or one month after yoga intervention finish).
  This concept was measured by a tool the Brief Health status Survey that was commonly used by nurses and doctors at Jumpandang Baru medical center to assess patients who are visiting the clinic. This tool has been shortened for the purpose of this study. The items include: (1) self-reported rating of their health status (ranging from 1: very poor to 6: excellent); (2) blood pressure (mmHg); (3) height (cm) and weight (kg) will be combined for calculating BMI; (4) stress in the past month; (5) smoking; (6) alcohol and illicit drug use and the percentage with which they use it to cope with stress; (7) prescription medication and over the counter medications for coping with stress, and the percentage with which they use it to cope with stress. Validity test will be performed before data collection begin. The brief health status survey will be performed in three different time to see how the yoga intervention change the health status of participants before and after intervention.
Coping Self-Efficacy Scale (The definition of coping self-efficacy is defined based on the concept proposed by Chesney et al in 2006 where they defined coping self-efficacy refers to the capacity to cope effectively with life obstacles. | (1) Pre-test (before yoga intervention), (2) Post-test one / at the week-eight (after yoga intervention finish), (3) Post-test two for following up (at the week twelve or one month after yoga intervention finish).
  The concept of coping self-efficacy is measured by the 26-item Coping Self-Efficacy Scale (CSES) developed by Chesney et. al (2006). Participants respond using an 11-point rating scale - 0 to 10, with anchor points on the scale at 0, meaning, 'I cannot do it at all'; 5, meaning, 'I am moderately certain I can do it'; and 10, meaning 'I am certain I can do it. This scale has good reliability with Cronbach's alpha for factor one (use problem-focused coping) was 0.91, factor two (stop unpleasant thought) was 0.91 and factor three (get support from family and friends) was 0.80 (Chesney et al., 2006). The coping self-efficacy scale will be performed in three different time to see how the yoga intervention change the coping self-efficacy level of participants before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Yen Chen, RN, PhD, Study Chair — National Taipei University of Nursing and Health Sciences; Jufri Hidayat, PhD (Cand), Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Jumpandang Baru Primary Health Care Center, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared under permission and with reasonable reason.

REFERENCES:
- [Result] Chesney MA, Neilands TB, Chambers DB, Taylor JM, Folkman S. A validity and reliability study of the coping self-efficacy scale. Br J Health Psychol. 2006 Sep;11(Pt 3):421-37. doi: 10.1348/135910705X53155. PMID 16870053
- [Result] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT05503680/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT05503680/ICF_001.pdf